CLINICAL TRIAL: NCT05412069
Title: A Multicenter, Prospective, Non-randomized Study on Pathophysiology, Diagnosis, and Biofeedback Therapy in Fecal Incontinence (FI) Using Fecobionics (NORMAL and ABNORMAL-FI)
Brief Title: Trial to Evaluate Fecobionics in Fecal Incontinence (FI) (NORMAL and ABNORMAL-FI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The California Medical Innovations Institute, Inc. (Other)
Collaborators: Augusta University Medical Center (Unknown)
Responsible Party: Principal Investigator, Hans Gregersen, PhD, Research Professor, The California Medical Innovations Institute, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CALM-CLIN-2022 new
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Normal Subjects; Fecal Incontinence
Keywords: anorectal; Fecobionics; defecation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecobionics study (Experimental): Fecobionics
  Interventions: Device: Fecobionics
- Feco BFT (Active Comparator): In this ARM Fecobionics will be used as a BFT tool
  Interventions: Device: Fecobionics

INTERVENTIONS:
Device: Fecobionics — Fecobionics is a novel device to be inserted through the anal canal into rectum for studying defecation. Anorectal manometry, balloon expulsion test, and anal ultrasonography will be used as reference.
  Other Names: anorectal manometry; balloon expulsion test; anal ultrasonography

SUMMARY:
The objective is to determine the length-tension properties of the anal sphincters using Fecobionics in normal subjects and FI patients during anal distension and during simulated evacuation. Fecobionics has the consistency and shape of normal stool and can record pressures, cross-sectional area, orientation and viscoelastic properties of the anorectum and can map the geometric profiles during evacuation, and thereby provides multi-dimensional measurements of pressures, deformability, and topographic changes. Fecobionics combines several existing tests to provide novel insight into anorectal function. The purpose for the development was to overcome the technological controversies and disagreement between various tests and unphysiological test conditions. The aim was to imitate defecation as much as possible to the natural process. Fecobionics was developed to simulate stool and to provide the driving pressure and resulting deformations of stool along with a measure of an objective anorectal angle during defecation in a single examination. Fecobionics makes it possible to describe objectively, without disturbing the defecation process, the opening characteristics and pressure signatures during initial entry into the relaxing anal canal.

The overall goal is to provide mechanistic understanding of defecation in health and defecatory disorders. It exceeds previous attempts to make artificial stool for evaluation of defecation (BET and FECOM) and integrates other technologies as well. It was designed to have a consistency and deformability of Type 4 (range type 3-5) on the Bristol stool form scale. The range from types 3-5 is found in 70% of normal subjects. A major novelty is that Fecobionics measures pressures in axial direction; i.e., in the flow direction.

DETAILED DESCRIPTION:
Defecatory disorders affect 25% of the population and the incidence is rising. These diseases pose a major health care burden and are poorly recognized and treated. The need for better diagnostics and therapeutics is substantial. Defecatory disorders including constipation and fecal incontinence are associated with diet, aging and a variety of underlying factors and diseases.

Current diagnostic tests such as the balloon expulsion test (BET), high-resolution anorectal manometry (HRM), defecography, and dynamic pelvic MRI are indirect surrogates for the act of defecation, and provide incomplete and often conflicting information, because most of them are not simulating defecation. Most tests are done with the subjects in lateral lying position, which is an abnormal posture for defecation. The results of these tests correlate poorly with symptoms and treatment outcomes. The simplest anorectal physiology test is the BET where a rectal balloon is filled with 50 ml water where expulsion within 1-2 min is considered normal. Anorectal manometry records the pressure exerted by the anal sphincters and puborectalis during rest and contraction. Defecography shows how well the rectum holds and evacuates the stool. Defecography uses a liquid with mechanical properties that are quite dissimilar to feces and hence cannot represent the physiology of defecation. Current research paradigms for defecatory disorders need a new technology that can provide real time, quantitative, and mechanistic insights by simulating defecation physiologically through multi-dimensional measurements of the pressure profiles, deformability, and topographic changes. The investigators have developed a wired Fecobionics device that integrates current tests to provide detailed mapping of physiological parameters during defecation of the device. This device has been further developed to a wireless device with expanded measurements. This was tested in the NORMAL study.

In this study, the investigators would like to learn more about FI patients and obtain ultrasonography data from 15 normal subjects for comparison. Fecal incontinence is a common problem, often nor properly diagnosed and treated. The goals are to determine the role of anorectal muscles in maintaining continence and defecation, and how their malfunction(s) can cause FI by using the new technology (i.e., Fecobionics) and novel methodology. Specifically, the investigators wish to determine the anal length-tension properties, a measure of the active and passive properties of the anal sphincter muscles, i.e. the compliance or stiffness.

Fecal incontinence (FI) affects 1 in 7 Americans with a rising incidence that poses a major healthcare burden. FI pathophysiology is poorly understood and consequently there is a dearth of effective treatment(s) compared to other defecatory disorders including constipation. A critical barrier to progress has been the lack of comprehensive, physiologically relevant and practical diagnostic test for identifying underlying mechanism(s). Current tests provide either incomplete or conflicting information that do not correlate with symptoms and treatment outcomes. The objective is to determine the role of anorectal muscles in maintaining continence and facilitating defecation, and how their malfunction(s) can cause FI by using a novel technology called Fecobionics (an electronic simulated stool) to evaluate the diagnostic and therapeutic utility of the novel technology. Fecobionics has the consistency and shape of normal stool and can record pressures, cross-sectional area, orientation and viscoelastic properties of the anorectum and can map the geometric profiles during evacuation, and thereby provides multi-dimensional measurements of pressures, deformability, and topographic changes. The central hypothesis is that the movement of the Fecobionics device through the anorectum will provide unknown and new mechanistic insights on anorectal physiology including length-tension properties of anorectal muscles, intraluminal pressure changes, deformability, and resistance generated during its movement and distensibility of the anal sphincters in NS and FI patients. Fecobionics studies have been done on more than 100 normal subjects and patients with anorectal disorders in Hong Kong using a structurally similar but simplified wired device that merely measured pressures. The published Fecobionics studies revealed clear differences between normal subjects and FI patients, as well as they demonstrated that the correlation with symptoms are higher with Fecobionics than with current technology (HRM-BET) and the outcome of biofeedback therapy can be predicted with Fecobionics. In this study, the Fecobionics upgraded hardware, software and graphical user interface (GUI) will be used to generate clinical data in FI patients and in later stages it will be used to guide biofeedback training (BT) in FI patients. Whether specific muscle length-tension properties, i.e., the relationship between muscle length and the force the anorectal muscle produces at that length, play a role in the evacuation and continence mechanics in NS and FI patients has not been studied in detail, and until now an appropriate method and system for such an analysis has not been available. The approach is based on promising data using 1) Anal EndoFLIP, 2) the previous wired Fecobionics prototype device (both invented by the PI) and 3) 3D ultrasound with vaginal distension for determining puborectalis length-tension properties, all of which have suggested that these properties are important. The overall objective is to validate a fully integrative dynamic investigational tool that mimics a normal stool for diagnostics and FI treatment. The expected outcomes are that the device will provide new mechanistic insights on anorectal physiology including the contributions of muscle length-tension properties, and facilitate development of new FI treatment strategies including improvement of BT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent;
2. Willing and able to undergo required study tests, surveys, and procedures;
3. Age > 18 years of age.

Exclusion Criteria:

1. Female who is pregnant;
2. Prior anorectal surgery;
3. Prior bowel resection;
4. History of chronic constipation;
5. In the opinion of the investigator, the subject is not a suitable candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Length-tension properties of the anal sphincter will be reported | 1.5 year
Front-rear pressure difference (in cmH2O) will be measured | 1.5 year
  Fecobionics contain pressure sensors in front end and rear end which can measure pressures

SECONDARY OUTCOMES:
Anorectal angle (in degree) will be measured | 1.5 year
  Fecobionics contain motion processing units with gyroscopes and accelerometers, which can measure angles
Expulsion velocity (in mm/s) will be reported | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gregersen, MD, PhD, Principal Investigator — California Medical Innovations Institute
Locations (2):
- United States (2):
  - California Medical Innovations Institute, San Diego, California
  - Augusta University Medical Center, Augusta, Georgia

IPD SHARING:
Plan to Share IPD: No